CLINICAL TRIAL: NCT00847665
Title: Comparison of Two Turning Regimens (2 Versus Every 4 Hours) in the Prevention of Pressure Ulcers in Patients on Mechanical Ventilation That Use Alternating-pressure Air Mattresses.
Brief Title: Pressure Ulcer Prevention in Ventilated Patients Using Two Repositioning Regimens
Acronym: PUPPAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Virgen de las Nieves (Other)
Responsible Party: Principal Investigator, Francisco Manzano Manzano, MD,PhD, University Hospital Virgen de las Nieves
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HVN-2308-2008
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Results first posted 2013-04-17 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-03

CONDITIONS: Pressure Ulcers
Keywords: Pressure ulcers; Repositioning; Prevention; Mechanical Ventilation; Critical care
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Turning every 4 hours (Active Comparator): The four-hours repositioning group patients were turned every four hours following the next sequence: left side, back with a 30º elevation of the head end and the foot end of the bed, right side using the 30º tilt, back.
  Interventions: Other: repositioning
- Turning every 2 hours (Experimental): The two-hours repositioning group patients, were turned every two hours following the next sequence: left side, back with a 30º elevation of the head end and the foot end of the bed, right side using the 30º tilt, back.
  Interventions: Other: repositioning

INTERVENTIONS:
Other: repositioning — Turning every 4 or 2 hours

SUMMARY:
The purpose of this study is to compare a 2-hour versus every 4-hour turning regimen on the incidence of grade > II pressure ulcers (PU) in patients in ICU on mechanical ventilation ≥ 24h that use alternating-pressure air mattresses (APAMs).

DETAILED DESCRIPTION:
Pressure ulcers (PUs) pose a major healthcare challenge and are associated with an increased risk of infection and sepsis, longer hospital stay, and higher hospitalization costs. Their reported incidence in critical care patients varies widely from 1% to 56%. Therefore it is important to take appropriate preventive measures, which can often be successful and less costly than the treatment of established ulcers. Among these measures are the use of pressure-reducing surfaces and repositioning strategies in a protocolized way. Though there is general agreement that critical care patients, including those under mechanical ventilation must use pressure-reducing surfaces, there is no enough evidence in the literature about what is the best repositioning schedule when new, high technology mattresses are used. The use of this new technology has lead to propose that repositioning can be less frequent. In the only clinical trial where this subject (time interval turning) has been addressed (Vanderwee et al, Journal of Advanced Nursing), it is concluded that a turning regimen every 4 hours is equally effective than a 2-hour turning, using this kind of mattresses. Nonetheless this study is not made in critically ill patients, that have more risk factors for developing PUs, the reason we don´t share this findings and recommendations cannot be generalized.

The study hypothesis is that in patients using APAMs, a turning regimen every 2 hour compared to a 4-hour is most effective in the prevention of PUs and could be equally safe.

The objective of this study is to investigate the effect of postural turnings every 2 hours compared to every 4 hours on the incidence of grade > II pressure ulcers (PU) in patients in ICU on mechanical ventilation (MV) ≥ 24h that use alternating-pressure air mattresses (APAMs) The study is an open label, randomized, controlled clinical trial. The main variable is the incidence of Pus grade ≥ II. As secondary variables measures of efficacy and safety of patients will be registered. The study will take place in a 26 bed medical-surgical ICU with APAMs. Randomization will be done between 24h-48h from the beginning of MV. The final analysis will be by intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the medical-surgical ICU, requiring more than 24 hours of mechanical ventilation.
* Patients on alternating-pressure air mattresses.
* Patients or their legal representative able to provide written informed consent to participate in the study
* Patients whose weight are within the limits accepted by the mattresses (45-140 Kg)
* Over 18 years

Exclusion Criteria:

* Patients with pressure ulcer at ICU admission.
* Pregnant patients
* Patients in which informed consent is not obtained in the first 48 hours of mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2009-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Manzano, MD,PhD, Principal Investigator — University Hospital Virgen de las Nieves
Locations (1):
- Hospital Universitario Virgen de las Nieves, Granada, Granada, Spain

REFERENCES:
- [Background] Vanderwee K, Grypdonck MH, De Bacquer D, Defloor T. Effectiveness of turning with unequal time intervals on the incidence of pressure ulcer lesions. J Adv Nurs. 2007 Jan;57(1):59-68. doi: 10.1111/j.1365-2648.2006.04060.x. PMID 17184374
- [Background] Defloor T, De Bacquer D, Grypdonck MH. The effect of various combinations of turning and pressure reducing devices on the incidence of pressure ulcers. Int J Nurs Stud. 2005 Jan;42(1):37-46. doi: 10.1016/j.ijnurstu.2004.05.013. PMID 15582638
- [Background] Krapfl LA, Gray M. Does regular repositioning prevent pressure ulcers? J Wound Ostomy Continence Nurs. 2008 Nov-Dec;35(6):571-7. doi: 10.1097/01.WON.0000341469.33567.61. PMID 19018196
- See also: University Hospital Virgen de las Nieves — http://www.hvn.es

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A medical-surgical ICU of a university hospital. Patients were recruited from february 2009 to January 2011
Pre-assignment Details: A total of 512 patients with more than 24 hours of mechanical ventilation were screened. 55 patients were excluded because of the presence of pressure ulcer. Other 126 patients were excluded because of the presence of other exclusion criteria (age, pregnancy, refusal of consent,...)
Groups:
- Turning Every 4 Hours: Repositioning by the nursing staff every four hours (left side, back with a 30º elevation of the head end and the foot end of the bed, right side, back), using the 30º tilt
- Turning Every 2 Hours: Repositioning by the nursing staff every two hours (left side, back with a 30º elevation of the head end and the foot end of the bed, right side, back), using the 30º tilt
Period: Overall Study
Arm/Group | Turning Every 4 Hours | Turning Every 2 Hours
Started | 165 | 165
Completed | 164 | 165
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Turning Every 4 Hours | Turning Every 2 Hours | Total
Number analyzed (Participants) | 165 | 165 | 330
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 89 | 81 | 170
  >=65 years | 76 | 84 | 160
Age Continuous [Mean (Standard Deviation); unit: years] | 61 (15) | 62 (14) | 61 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 56 | 110
  Male | 111 | 109 | 220
Region of Enrollment [Number; unit: participants]
  Spain | 165 | 165 | 330

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Pressure Ulcer (PU) Grade ≥ II
Description: Pressure ulcers were categorized according to the EPUAP-classification system. A grade I PU is non-blanchable erythema, a grade II is an abrasion or blister, a grade III is a superficial ulcer and a grade IV is a deep ulcer
Time Frame: Intensive Care Unit (ICU) length of stay (days)
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Turning Every 4 Hours | Turning Every 2 Hours
Number analyzed (Participants) | 164 | 165
participants | 22 | 17

2. Secondary Outcome: ICU Mortality
Description: ICU mortality (number of death in ICU)
Time Frame: ICU length of stay (an average of 28 days)
Measure: Number; unit: participants
Arm/Group | Turning Every 4 Hours | Turning Every 2 Hours
Number analyzed (Participants) | 164 | 165
participants | 51 | 60

3. Secondary Outcome: Workload of Nurses
Description: Time actually spent to manual repositioning by nurses team, in minutes/day
Time Frame: icu length of stay
Measure: Median (Inter-Quartile Range); unit: minutes per day
Arm/Group | Turning Every 4 Hours | Turning Every 2 Hours
Number analyzed (Participants) | 164 | 165
minutes per day | 10.6 [7.9 to 14.9] | 20.8 [14.4 to 27.4]

4. Secondary Outcome: Length of Mechanical Ventilation (MV)
Description: Time from initiation to withdrawal of mechanical ventilation. Days
Time Frame: ICU length of stay
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Turning Every 4 Hours | Turning Every 2 Hours
Number analyzed (Participants) | 164 | 165
days | 8 [5 to 15] | 7 [3 to 15]

ADVERSE EVENTS:
Time Frame: 2 year
Description: ICU length of stay for each patient
Arm/Group | Turning Every 4 Hours | Turning Every 2 Hours
Serious Adverse Events (participants affected / at risk) | 15/164 | 23/165
Other Adverse Events (participants affected / at risk) | 50/164 | 60/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Turning Every 4 Hours (N=164) | Turning Every 2 Hours (N=165)
unplanned extubation (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 19 (19) — Unplanned extubation is defined as premature removal of the endotracheal tube by action of the patient or during care and manipulation of the patient
Loss of medical devices (Surgical and medical procedures) | 12 (12) | 15 (15)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Turning Every 4 Hours (N=164) | Turning Every 2 Hours (N=165)
Endotracheal tube obstruction (Respiratory, thoracic and mediastinal disorders) | 50 (50) | 60 (60) — Defined when clinically suspected and diagnosed by the attended physician, because of the presence of visible airway secretion into the endotracheal tube. There was always the need to use isotonic saline instillation before tracheal suctioning.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No